CLINICAL TRIAL: NCT01765335
Title: Heart Failure Re-admission Risk Estimation Using NICaS System With Comparison to Serum BNP Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of R&D, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NICaS CHF
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure
Keywords: heart failure, BNP, NICaS system, readmition
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NICaS system efficacy in HF patients (Experimental): NICaS system efficacy in HF patients
  Interventions: Device: NICaS system

INTERVENTIONS:
Device: NICaS system — NICaS parameters (cardiac output and total peripheral resistance) and serum BNP levels will be processed in an excel sheet including study reference number to keep confidentiality

SUMMARY:
HF represents a major burden in the developed world. Mortality and rehospitalization rates post-discharge in patients admitted with HF may be as high as 15%-30% within 60-90 days, respectively. Given that rehospitalization drives much of the cost associated with HF, there has been increased interest in predicting risk of rehospitalization as a means to control health care costs. These risk stratification models can serve as important clinical tools by helping to identify those patients who are at very high risk may be observed more closely or treated more intensively. The most important predictors for the combined endpoint of death or rehospitalization were admission serum creatinine concentration, systolic blood pressure,admission hemoglobin level, discharge use of ACE-Ior ARBS, and Pulmonary disease. Other independent predictors during hospitalization of readmission and mortality included low admission Kansas City Cardiomyopathy Questionnaire score, high BNP, hyponatremia, tachycardia, hypotension, absence of b-blocker therapy, and history of diabetes and arrhythmias. Nevertheless, both models fail to provide the treating physician a simple decision making tool for predicting which patient is stable enough to be discharged from the hospital without a high risk of readmission. The Non Invasive Cardiac System (NICaS, Israel), calculates the cardiac output by measuring impedance cardiography in a tetra-polar mode, derived from electrodes placed on both wrists or one wrist and the contra-lateral ankle. This simple to operate, non-invasive technique was validated in a few studies to be reliable in estimation of CO compared to traditional, invasive techniques in different settings including HF patients. A previous study demonstrated that parameters derived from this system showed a highly significant correlation to echo estimated EF and serum BNP in chronic HF patients and were equally able to predict complications in this population. Aim:To assess whether the NICaS system can identify high risk HF patient for readmission prior to their discharge compared to serum BNP measurement.

DETAILED DESCRIPTION:
Heart failure represents a major burden in the developed world. Mortality and rehospitalization rates post-discharge in patients admitted with HF may be as high as 15% and 30% within 60-90 days, respectively. Given that rehospitalization drives much of the cost associated with HF, there has been increased interest in predicting risk of rehospitalization as a means to control health care costs. These risk stratification models can serve as important clinical tools by helping to identify those patients who are at very high risk may be observed more closely or treated more intensively. The most important predictors for the combined endpoint of death or rehospitalization were admission serum creatinine concentration, systolic blood pressure,admission hemoglobin level, discharge use of ACE-Ior ARBS, and Pulmonary disease. Other independent predictors during hospitalization of readmission and mortality included low admission Kansas City Cardiomyopathy Questionnaire score, high BNP, hyponatremia, tachycardia, hypotension, absence of b-blocker therapy, and history of diabetes and arrhythmias. Nevertheless, both models fail to provide the treating physician a simple decision making tool for predicting which patient is stable enough to be discharged from the hospital without a high risk of readmission. The Non Invasive Cardiac System (NICaS, Israel), calculates the cardiac output by measuring impedance cardiography in a tetra-polar mode, derived from electrodes placed on both wrists or one wrist and the contra-lateral ankle. This simple to operate, non-invasive technique was validated in a few studies to be reliable in estimation of CO compared to traditional, invasive techniques in different settings including HF patients. A previous study demonstrated that parameters derived from this system showed a highly significant correlation to echo estimated EF and serum BNP in chronic HF patients and were equally able to predict complications in this population. Aim:To assess whether the NICaS system can identify high risk HF patient for readmission prior to their discharge compared to serum BNP measurement.Methods and population:Known HF patients, admitted due to HF exacerbation, will be tested with NICaS system in concordance with serum BNP measurement prior to their discharge from the hospital. The decision for discharge will be made on clinical ground by the treating physician alone. The patients will be tested by NICaS system in the following manner-patches will be attached to both patient's wrists, or one wrist and contra-lateral ankle for a period of approximately 30 seconds. During that time the patient will be seated or supine.3cc of blood will be drawn from peripheral vein for BNP level measurement.NICaS parameters and serum BNP levels will be processed in an excel sheet. The patients will be followed by a telephone questionnaire after 3 months from discharge in order to document events of readmission or death.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. HF admitted patient from cardiology and internal medicine departments in our institution.

Exclusion Criteria:

1. Severe aortic valve regurgitation and/or aortic stenosis.
2. Aortic aneurysm.
3. Heart rate above 130 beats/min.
4. Intra- and extra-cardiac shunts.
5. Severe peripheral vascular disease.
6. Severe pitting edema.
7. Sepsis.
8. Use of hemodialysis.
9. Patients under 18 years of age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
HF readmition | 3 months
  To assess whether the NICaS system can identify high risk HF patient for readmission prior to their discharge compared to serum BNP measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Havakuk, MD, Study Director — Tel Aviv Medical Center
Locations (1):
- Tel Aviv SoUrasky MC, Tel Aviv, Israel